CLINICAL TRIAL: NCT04646200
Title: Cognitive Behavioral Therapy For Insomnia (CBT-I) to Improve Functional Outcomes in Veterans With Psychosis
Brief Title: CBT-I to Improve Functional Outcomes in Veterans With Psychosis
Acronym: CBT-I Merit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3213-R; I01RX003213 (NIH)
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Insomnia; Psychosis
Keywords: Mental Disorders; Insomnia Disorder; Psychosis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychotic Disorders; Mental Disorders | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy-Insomnia (Experimental): CBT-I addresses cognitive, arousal and behavioral factors related to sleep difficulties. Sessions combine assessment, conceptualization, psychoeducation, behavioral strategies and cognitive therapy, using a consistent structure including review of participants' sleep log and adherence to behavioral guidelines, modification of time in bed, cognitive therapy, and relaxation techniques. CBT-I also incorporates psychoeducation about biological and psychological elements that regulate sleep. Other strategies include stimulus control (i.e., getting out of bed when not sleepy) to extinguish the conditioned arousal common in insomnia, and relaxation techniques to reduce arousal associated with the bed, bedroom, or bedtime.
  Interventions: Behavioral: Cognitive Behavioral Therapy-Insomnia
- Health and Wellness (Active Comparator): Health and Wellness is a general self-management curriculum focused on providing education and support for managing physical and emotional well-being. Each session follows a basic structure including review of previous session material, new educational information and discussion on several topics over the course of single or multiple sessions. Each session will focus on the impact of the topic on overall health and wellness, identifying benefits and challenges to improving or maintaining health in that area, and strategies that clients may find helpful to address challenges in that area. Example topics include physical activity/exercise, nutrition/healthy eating, managing medications and side effects, and addictive behaviors (e.g., substance use, gambling, eating).
  Interventions: Behavioral: Health and Wellness

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy-Insomnia — CBT-I addresses cognitive, arousal and behavioral factors related to sleep difficulties. Sessions combine assessment, conceptualization, psychoeducation, behavioral strategies and cognitive therapy, using a consistent structure including review of participants' sleep log and adherence to behavioral guidelines, modification of time in bed, cognitive therapy, and relaxation techniques. CBT-I also incorporates psychoeducation about biological and psychological elements that regulate sleep. Other strategies include stimulus control (i.e., getting out of bed when not sleepy) to extinguish the conditioned arousal common in insomnia, and relaxation techniques to reduce arousal associated with the bed, bedroom, or bedtime.
  Arms: Cognitive Behavioral Therapy-Insomnia
Behavioral: Health and Wellness — Health and Wellness is a general self-management curriculum focused on providing education and support for managing physical and emotional well-being. Each session follows a basic structure including review of previous session material, new educational information and discussion on several topics over the course of single or multiple sessions. Each session will focus on the impact of the topic on overall health and wellness, identifying benefits and challenges to improving or maintaining health in that area, and strategies that clients may find helpful to address challenges in that area. Example topics include physical activity/exercise, nutrition/healthy eating, managing medications and side effects, and addictive behaviors (e.g., substance use, gambling, eating).
  Arms: Health and Wellness

SUMMARY:
The goal of this project is to examine the efficacy of Cognitive Behavioral Therapy for Insomnia (CBT-I) for improving sleep and related functional outcomes in Veterans with psychosis and insomnia.

DETAILED DESCRIPTION:
The goal of this project is to examine the efficacy of Cognitive Behavioral Therapy for Insomnia (CBT-I) for improving sleep and related functional outcomes in Veterans with psychosis and insomnia.

Aim 1: Evaluate the efficacy of CBT-I for reducing insomnia severity in Veterans with psychosis and insomnia.

Hypothesis 1: CBT-I participants, as compared to those in an active control condition, will show significantly greater reductions on the Insomnia Severity Index at post-treatment and at a 6-month follow-up.

Aim 2: Evaluate the efficacy of CBT-I for improving the functioning of Veterans with psychosis and insomnia. Hypothesis 2: CBT-I participants, as compared to those in an active control condition, will show significantly greater increases in mental and physical health functioning on the Veterans RAND 36-Item Health Survey at post-treatment and at a 6-month follow-up.

Aim 3: Evaluate the process that underlies the relationship between insomnia severity and functioning in Veterans with psychosis and insomnia.

Hypothesis 3: The effect of CBT-I on mental and physical health functioning at post-treatment will be mediated by reductions in insomnia severity at week 5 of treatment.

Hypothesis 4: The effect of CBT-I on mental and physical health functioning at the 6-month follow-up will be mediated by reductions in insomnia severity at immediate post-treatment.

Exploratory Aim: Explore whether psychiatric symptoms 1) moderate the impact of CBT-I on insomnia and functioning and/or 2) change as a result of participation in CBT-I.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for SMI: Schizophrenic disorder, affective psychosis, major depression with psychotic features, delusional disorder, brief psychotic disorder, unspecified psychotic disorder, schizotypal personality disorder
* be between the ages of 18 and 80
* be actively participating in outpatient mental health services at designated site

Exclusion Criteria:

* currently in CBT-I treatment
* planning to move out of the area during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Participants will be assessed following completion of the study intervention, an expected average of 12 weeks; and again after approximately 6 months.
  Change in the ISI score; higher scores signify greater insomnia severity; scores range from 0 to 28.
Veterans RAND 36-item Health Survey (VR-36) | Participants will be assessed following completion of the study intervention, an expected average of 12 weeks; and again after approximately 6 months.
  Change in the VR-36 score; higher scores signify a more favorable health state; scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Klingaman, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No